CLINICAL TRIAL: NCT01239199
Title: Is the Exhaled Nitric Oxide in Infants a Predictive Marker of Asthma?
Brief Title: Is the Exhaled Nitric Oxide in Infants a Predictive Marker of Asthma ?
Acronym: NOnourisson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P 070802
Record Dates: First submitted 2010-10-21; First posted 2010-11-11 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Asthma
Keywords: Infants; Exhaled Nitric Oxide; Asthma; Tobacco smoke exposure; environment
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exhaled NO (Experimental)
  Interventions: Other: Measure of the exhaled NO

INTERVENTIONS:
Other: Measure of the exhaled NO — The exhaled NO will be measure by chemiluminescence in current ventilation by an indirect method (off-line)

SUMMARY:
Background:

It seems that in the infants and the young children, the increase of the Exhaled Nitric Oxide (eNO) is in connection with: (1) the risk of developing respiratory symptoms; (2) the risk of family and personal atopy; (3) the intensity of the respiratory symptoms; (4) the risk of passage of recurrent wheezing to asthma; (5) and contrary to the fact that the investigators noticed at the child's a positive relation with the environmental tobacco smoke

Objective: the investigators objective is to bring to light that the rise of the eNO, a non invasive biomarker of the bronchial inflammation, would be a risk factor expected from passage of recurrent wheezing of the infant and the young child (of less than 36 months old) towards the asthma of the child.Methods: Once the diagnosis of recurrent wheezing established, the investigators estimate by questionnaire the severity of the asthma, the personal and familial atopy, the collection of the environmental data. After allergic exploration (skin tests and assay of serum total and specific IgE, complete blood count), the eNO is measured by an off-line tidal breathing method using a chemiluminescence NO analyzer. Annually, a questionnaire will be send to families to appreciate the persistence or the remission of the asthma. After a simple descriptive analysis of the population and a multifactorial descriptive analysis, the investigators shall look for the connections between the rise of the eNO and the various clinical, biological and environmental parameters known to influence the variations of this marker. Then the investigators shall select a set of explanatory variables for a multivariate analysis by a logistic regression step by step.

DETAILED DESCRIPTION:
This study is a epidemiological observation study

ELIGIBILITY:
Inclusion Criteria:

* Infant between 6 and 36 months
* More than 3 wheezing episodes
* Questionary and biological assessment for recurrent wheeze
* Signature of the consent by 2 parents or by the only one of 2 parents (if this last one is the only present in the inclusion of the child)

Exclusion Criteria:

* Infant with respiratory disease in neonatal period
* Infant with other obstructive pathology (cystic fibrosis, Primary Ciliary Dyskinesia,…)
* Infant who have a respiratory infection less than 4 weeks
* Infant with asthma exacerbation or who still have corticosteroid treatment
* Infant without social security from their parents

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Measure of exhaled nitric oxide at the beginning of the study and incidence of asthma symptoms after 3 years of follow up | 1 day

SECONDARY OUTCOMES:
Atopic status with total and specific IgE levels and skin test, complete blood count | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Just, Principal Investigator — Trousseau Hospital - APHP
Locations (1):
- Service of multidisciplinary paediatrics (Armand-Trousseau Hospital), Paris, Île-de-France Region, France

REFERENCES:
- [Background] Lowe L, Custovic A, Woodcock A. Childhood asthma. Curr Allergy Asthma Rep. 2004 Mar;4(2):159-65. doi: 10.1007/s11882-004-0062-9. PMID 14769266
- [Background] Saglani S, Nicholson AG, Scallan M, Balfour-Lynn I, Rosenthal M, Payne DN, Bush A. Investigation of young children with severe recurrent wheeze: any clinical benefit? Eur Respir J. 2006 Jan;27(1):29-35. doi: 10.1183/09031936.06.00030605. PMID 16387932
- [Background] Pohunek P, Warner JO, Turzikova J, Kudrmann J, Roche WR. Markers of eosinophilic inflammation and tissue re-modelling in children before clinically diagnosed bronchial asthma. Pediatr Allergy Immunol. 2005 Feb;16(1):43-51. doi: 10.1111/j.1399-3038.2005.00239.x. PMID 15693911
- [Background] Franklin PJ, Turner SW, Mutch RC, Stick SM. Comparison of single-breath and tidal breathing exhaled nitric oxide levels in infants. Eur Respir J. 2004 Mar;23(3):369-72. doi: 10.1183/09031936.04.00084604. PMID 15065823
- [Background] Yang H, Wei W, Menconi M, Hasselgren PO. Dexamethasone-induced protein degradation in cultured myotubes is p300/HAT dependent. Am J Physiol Regul Integr Comp Physiol. 2007 Jan;292(1):R337-4. doi: 10.1152/ajpregu.00230.2006. Epub 2006 Sep 14. PMID 16973938
- [Background] Baraldi E, Dario C, Ongaro R, Scollo M, Azzolin NM, Panza N, Paganini N, Zacchello F. Exhaled nitric oxide concentrations during treatment of wheezing exacerbation in infants and young children. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1284-8. doi: 10.1164/ajrccm.159.4.9807084. PMID 10194178
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Background] Phelan PD, Robertson CF, Olinsky A. The Melbourne Asthma Study: 1964-1999. J Allergy Clin Immunol. 2002 Feb;109(2):189-94. doi: 10.1067/mai.2002.120951. PMID 11842286
- [Background] Zeiger RS, Dawson C, Weiss S. Relationships between duration of asthma and asthma severity among children in the Childhood Asthma Management Program (CAMP). J Allergy Clin Immunol. 1999 Mar;103(3 Pt 1):376-87. doi: 10.1016/s0091-6749(99)70460-4. PMID 10069869
- [Background] Harris JR, Magnus P, Samuelsen SO, Tambs K. No evidence for effects of family environment on asthma. A retrospective study of Norwegian twins. Am J Respir Crit Care Med. 1997 Jul;156(1):43-9. doi: 10.1164/ajrccm.156.1.9609094. PMID 9230724
- [Background] Martinez FD, Wright AL, Taussig LM, Holberg CJ, Halonen M, Morgan WJ. Asthma and wheezing in the first six years of life. The Group Health Medical Associates. N Engl J Med. 1995 Jan 19;332(3):133-8. doi: 10.1056/NEJM199501193320301. PMID 7800004
- [Background] Young S, Le Souef PN, Geelhoed GC, Stick SM, Turner KJ, Landau LI. The influence of a family history of asthma and parental smoking on airway responsiveness in early infancy. N Engl J Med. 1991 Apr 25;324(17):1168-73. doi: 10.1056/NEJM199104253241704. PMID 2011160
- [Background] Murray CS, Pipis SD, McArdle EC, Lowe LA, Custovic A, Woodcock A; National Asthma Campaign-Manchester Asthma and Allergy Study Group. Lung function at one month of age as a risk factor for infant respiratory symptoms in a high risk population. Thorax. 2002 May;57(5):388-92. doi: 10.1136/thorax.57.5.388. PMID 11978912
- [Background] Wahn U, Lau S, Bergmann R, Kulig M, Forster J, Bergmann K, Bauer CP, Guggenmoos-Holzmann I. Indoor allergen exposure is a risk factor for sensitization during the first three years of life. J Allergy Clin Immunol. 1997 Jun;99(6 Pt 1):763-9. doi: 10.1016/s0091-6749(97)80009-7. PMID 9215243
- [Background] Sears MR, Herbison GP, Holdaway MD, Hewitt CJ, Flannery EM, Silva PA. The relative risks of sensitivity to grass pollen, house dust mite and cat dander in the development of childhood asthma. Clin Exp Allergy. 1989 Jul;19(4):419-24. doi: 10.1111/j.1365-2222.1989.tb02408.x. PMID 2758355
- [Background] Lowe L, Murray CS, Custovic A, Simpson BM, Kissen PM, Woodcock A; NAC Manchester Asthma and Allergy Study Group. Specific airway resistance in 3-year-old children: a prospective cohort study. Lancet. 2002 Jun 1;359(9321):1904-8. doi: 10.1016/S0140-6736(02)08781-0. PMID 12057553
- [Background] Illi S, von Mutius E, Lau S, Niggemann B, Gruber C, Wahn U; Multicentre Allergy Study (MAS) group. Perennial allergen sensitisation early in life and chronic asthma in children: a birth cohort study. Lancet. 2006 Aug 26;368(9537):763-70. doi: 10.1016/S0140-6736(06)69286-6. PMID 16935687
- [Background] Strachan DP. Hay fever, hygiene, and household size. BMJ. 1989 Nov 18;299(6710):1259-60. doi: 10.1136/bmj.299.6710.1259. No abstract available. PMID 2513902
- [Background] Celedon JC, Wright RJ, Litonjua AA, Sredl D, Ryan L, Weiss ST, Gold DR. Day care attendance in early life, maternal history of asthma, and asthma at the age of 6 years. Am J Respir Crit Care Med. 2003 May 1;167(9):1239-43. doi: 10.1164/rccm.200209-1063OC. Epub 2002 Nov 21. PMID 12446273
- [Background] Braun-Fahrlander C, Gassner M, Grize L, Neu U, Sennhauser FH, Varonier HS, Vuille JC, Wuthrich B. Prevalence of hay fever and allergic sensitization in farmer's children and their peers living in the same rural community. SCARPOL team. Swiss Study on Childhood Allergy and Respiratory Symptoms with Respect to Air Pollution. Clin Exp Allergy. 1999 Jan;29(1):28-34. doi: 10.1046/j.1365-2222.1999.00479.x. PMID 10051699
- [Background] von Mutius E. Environmental factors influencing the development and progression of pediatric asthma. J Allergy Clin Immunol. 2002 Jun;109(6 Suppl):S525-32. doi: 10.1067/mai.2002.124565. PMID 12063508
- [Background] Ownby DR, Johnson CC, Peterson EL. Exposure to dogs and cats in the first year of life and risk of allergic sensitization at 6 to 7 years of age. JAMA. 2002 Aug 28;288(8):963-72. doi: 10.1001/jama.288.8.963. PMID 12190366
- [Background] Sigurs N, Gustafsson PM, Bjarnason R, Lundberg F, Schmidt S, Sigurbergsson F, Kjellman B. Severe respiratory syncytial virus bronchiolitis in infancy and asthma and allergy at age 13. Am J Respir Crit Care Med. 2005 Jan 15;171(2):137-41. doi: 10.1164/rccm.200406-730OC. Epub 2004 Oct 29. PMID 15516534
- [Background] Renzi PM, Turgeon JP, Marcotte JE, Drblik SP, Berube D, Gagnon MF, Spier S. Reduced interferon-gamma production in infants with bronchiolitis and asthma. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1417-22. doi: 10.1164/ajrccm.159.5.9805080. PMID 10228104
- [Background] Castro-Rodriguez JA, Holberg CJ, Wright AL, Martinez FD. A clinical index to define risk of asthma in young children with recurrent wheezing. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1403-6. doi: 10.1164/ajrccm.162.4.9912111. PMID 11029352
- [Background] Guilbert TW, Morgan WJ, Zeiger RS, Mauger DT, Boehmer SJ, Szefler SJ, Bacharier LB, Lemanske RF Jr, Strunk RC, Allen DB, Bloomberg GR, Heldt G, Krawiec M, Larsen G, Liu AH, Chinchilli VM, Sorkness CA, Taussig LM, Martinez FD. Long-term inhaled corticosteroids in preschool children at high risk for asthma. N Engl J Med. 2006 May 11;354(19):1985-97. doi: 10.1056/NEJMoa051378. PMID 16687711
- [Background] Redington AE, Meng QH, Springall DR, Evans TJ, Creminon C, Maclouf J, Holgate ST, Howarth PH, Polak JM. Increased expression of inducible nitric oxide synthase and cyclo-oxygenase-2 in the airway epithelium of asthmatic subjects and regulation by corticosteroid treatment. Thorax. 2001 May;56(5):351-7. doi: 10.1136/thorax.56.5.351. PMID 11312402
- [Background] Asano K, Chee CB, Gaston B, Lilly CM, Gerard C, Drazen JM, Stamler JS. Constitutive and inducible nitric oxide synthase gene expression, regulation, and activity in human lung epithelial cells. Proc Natl Acad Sci U S A. 1994 Oct 11;91(21):10089-93. doi: 10.1073/pnas.91.21.10089. PMID 7524082
- [Background] Pijnenburg MW, Lissenberg ET, Hofhuis W, Ghiro L, Ho WC, Holland WP, de Jongste JC. Exhaled nitric oxide measurements with dynamic flow restriction in children aged 4-8 yrs. Eur Respir J. 2002 Oct;20(4):919-24. doi: 10.1183/09031936.02.01282002. PMID 12412684
- [Background] Murphy AW, Platts-Mills TA, Lobo M, Hayden F. Respiratory nitric oxide levels in experimental human influenza. Chest. 1998 Aug;114(2):452-6. doi: 10.1378/chest.114.2.452. PMID 9726729
- [Background] Ferreira IM, Hazari MS, Gutierrez C, Zamel N, Chapman KR. Exhaled nitric oxide and hydrogen peroxide in patients with chronic obstructive pulmonary disease: effects of inhaled beclomethasone. Am J Respir Crit Care Med. 2001 Sep 15;164(6):1012-5. doi: 10.1164/ajrccm.164.6.2012139. PMID 11587988
- [Background] Lindberg S, Cervin A, Runer T. Low levels of nasal nitric oxide (NO) correlate to impaired mucociliary function in the upper airways. Acta Otolaryngol. 1997 Sep;117(5):728-34. doi: 10.3109/00016489709113468. PMID 9349871
- [Background] Lundberg JO, Nordvall SL, Weitzberg E, Kollberg H, Alving K. Exhaled nitric oxide in paediatric asthma and cystic fibrosis. Arch Dis Child. 1996 Oct;75(4):323-6. doi: 10.1136/adc.75.4.323. PMID 8984919
- [Background] Frey U, Kuehni C, Roiha H, Cernelc M, Reinmann B, Wildhaber JH, Hall GL. Maternal atopic disease modifies effects of prenatal risk factors on exhaled nitric oxide in infants. Am J Respir Crit Care Med. 2004 Aug 1;170(3):260-5. doi: 10.1164/rccm.200307-1002OC. Epub 2004 Apr 1. PMID 15059789
- [Background] Kharitonov SA, Robbins RA, Yates D, Keatings V, Barnes PJ. Acute and chronic effects of cigarette smoking on exhaled nitric oxide. Am J Respir Crit Care Med. 1995 Aug;152(2):609-12. doi: 10.1164/ajrccm.152.2.7543345.
- [Background] Moncada S, Higgs A. The L-arginine-nitric oxide pathway. N Engl J Med. 1993 Dec 30;329(27):2002-12. doi: 10.1056/NEJM199312303292706. No abstract available. PMID 7504210
- [Background] Hamid Q, Springall DR, Riveros-Moreno V, Chanez P, Howarth P, Redington A, Bousquet J, Godard P, Holgate S, Polak JM. Induction of nitric oxide synthase in asthma. Lancet. 1993 Dec 18-25;342(8886-8887):1510-3. doi: 10.1016/s0140-6736(05)80083-2. PMID 7504773
- [Background] Franklin PJ, Taplin R, Stick SM. A community study of exhaled nitric oxide in healthy children. Am J Respir Crit Care Med. 1999 Jan;159(1):69-73. doi: 10.1164/ajrccm.159.1.9804134. PMID 9872820
- [Background] Gratziou C, Lignos M, Dassiou M, Roussos C. Influence of atopy on exhaled nitric oxide in patients with stable asthma and rhinitis. Eur Respir J. 1999 Oct;14(4):897-901. doi: 10.1034/j.1399-3003.1999.14d28.x. PMID 10573239
- [Background] Avital A, Uwyyed K, Berkman N, Bar-Yishay E, Godfrey S, Springer C. Exhaled nitric oxide is age-dependent in asthma. Pediatr Pulmonol. 2003 Nov;36(5):433-8. doi: 10.1002/ppul.10377. PMID 14520727
- [Background] Lanz MJ, Leung DY, McCormick DR, Harbeck R, Szefler SJ, White CW. Comparison of exhaled nitric oxide, serum eosinophilic cationic protein, and soluble interleukin-2 receptor in exacerbations of pediatric asthma. Pediatr Pulmonol. 1997 Nov;24(5):305-11. doi: 10.1002/(sici)1099-0496(199711)24:53.0.co;2-h. PMID 9407562
- [Background] Mahut B, Delclaux C, Tillie-Leblond I, Gosset P, Delacourt C, Zerah-Lancner F, Harf A, de Blic J. Both inflammation and remodeling influence nitric oxide output in children with refractory asthma. J Allergy Clin Immunol. 2004 Feb;113(2):252-6. doi: 10.1016/j.jaci.2003.10.038. PMID 14767438
- [Background] Silvestri M, Sabatini F, Spallarossa D, Fregonese L, Battistini E, Biraghi MG, Rossi GA. Exhaled nitric oxide levels in non-allergic and allergic mono- or polysensitised children with asthma. Thorax. 2001 Nov;56(11):857-62. doi: 10.1136/thorax.56.11.857. PMID 11641510
- [Background] Silvestri M, Sabatini F, Sale R, Defilippi AC, Fregonese L, Battistini E, Biraghi MG, Rossi GA. Correlations between exhaled nitric oxide levels, blood eosinophilia, and airway obstruction reversibility in childhood asthma are detectable only in atopic individuals. Pediatr Pulmonol. 2003 May;35(5):358-63. doi: 10.1002/ppul.10264. PMID 12687592
- [Background] Jouaville LF, Annesi-Maesano I, Nguyen LT, Bocage AS, Bedu M, Caillaud D. Interrelationships among asthma, atopy, rhinitis and exhaled nitric oxide in a population-based sample of children. Clin Exp Allergy. 2003 Nov;33(11):1506-11. doi: 10.1046/j.1365-2222.2003.01800.x. PMID 14616861
- [Background] Barreto M, Villa MP, Martella S, Ronchetti F, Darder MT, Falasca C, Pagani J, Massa F, Ronchetti R. Exhaled nitric oxide in asthmatic and non-asthmatic children: influence of type of allergen sensitization and exposure to tobacco smoke. Pediatr Allergy Immunol. 2001 Oct;12(5):247-56. doi: 10.1034/j.1399-3038.2001.00041.x. PMID 11737671
- [Background] Warke TJ, Fitch PS, Brown V, Taylor R, Lyons JD, Ennis M, Shields MD. Exhaled nitric oxide correlates with airway eosinophils in childhood asthma. Thorax. 2002 May;57(5):383-7. doi: 10.1136/thorax.57.5.383. PMID 11978911
- [Background] Bratton DL, Lanz MJ, Miyazawa N, White CW, Silkoff PE. Exhaled nitric oxide before and after montelukast sodium therapy in school-age children with chronic asthma: a preliminary study. Pediatr Pulmonol. 1999 Dec;28(6):402-7. doi: 10.1002/(sici)1099-0496(199912)28:63.0.co;2-v. PMID 10587413
- [Background] Di Rosa M, Radomski M, Carnuccio R, Moncada S. Glucocorticoids inhibit the induction of nitric oxide synthase in macrophages. Biochem Biophys Res Commun. 1990 Nov 15;172(3):1246-52. doi: 10.1016/0006-291x(90)91583-e. PMID 1700905
- [Background] Malmberg LP, Pelkonen AS, Haahtela T, Turpeinen M. Exhaled nitric oxide rather than lung function distinguishes preschool children with probable asthma. Thorax. 2003 Jun;58(6):494-9. doi: 10.1136/thorax.58.6.494. PMID 12775859
- [Background] Nathan C, Xie QW. Nitric oxide synthases: roles, tolls, and controls. Cell. 1994 Sep 23;78(6):915-8. doi: 10.1016/0092-8674(94)90266-6. No abstract available. PMID 7522969
- [Background] Thomas NS, Wilkinson J, Holgate ST. The candidate region approach to the genetics of asthma and allergy. Am J Respir Crit Care Med. 1997 Oct;156(4 Pt 2):S144-51. doi: 10.1164/ajrccm.156.4.12-tac-13. PMID 9351596
- [Background] Grasemann H, Yandava CN, Drazen JM. Neuronal NO synthase (NOS1) is a major candidate gene for asthma. Clin Exp Allergy. 1999 Dec;29 Suppl 4:39-41. PMID 10641565
- [Background] Grasemann H, Yandava CN, Storm van's Gravesande K, Deykin A, Pillari A, Ma J, Sonna LA, Lilly C, Stampfer MJ, Israel E, Silverman EK, Drazen JM. A neuronal NO synthase (NOS1) gene polymorphism is associated with asthma. Biochem Biophys Res Commun. 2000 Jun 7;272(2):391-4. doi: 10.1006/bbrc.2000.2794. PMID 10833424
- [Background] Wechsler ME, Grasemann H, Deykin A, Silverman EK, Yandava CN, Israel E, Wand M, Drazen JM. Exhaled nitric oxide in patients with asthma: association with NOS1 genotype. Am J Respir Crit Care Med. 2000 Dec;162(6):2043-7. doi: 10.1164/ajrccm.162.6.2003089. PMID 11112111
- [Background] Holla LI, Schuller M, Buckova D, Vacha J. Neuronal nitric oxide synthase gene polymorphism and IgE-mediated allergy in the Central European population. Allergy. 2004 May;59(5):548-52. doi: 10.1111/j.1398-9995.2004.00458.x. PMID 15080837
- [Background] Leung TF, Liu EK, Tang NL, Ko FW, Li CY, Lam CW, Wong GW. Nitric oxide synthase polymorphisms and asthma phenotypes in Chinese children. Clin Exp Allergy. 2005 Oct;35(10):1288-94. doi: 10.1111/j.1365-2222.2005.02342.x. PMID 16238787
- [Background] Lee YC, Cheon KT, Lee HB, Kim W, Rhee YK, Kim DS. Gene polymorphisms of endothelial nitric oxide synthase and angiotensin-converting enzyme in patients with asthma. Allergy. 2000 Oct;55(10):959-63. doi: 10.1034/j.1398-9995.2000.00724.x. PMID 11030378
- [Background] Holla LI, Buckova D, Kuhrova V, Stejskalova A, Francova H, Znojil V, Vacha J. Prevalence of endothelial nitric oxide synthase gene polymorphisms in patients with atopic asthma. Clin Exp Allergy. 2002 Aug;32(8):1193-8. doi: 10.1046/j.1365-2745.2002.01445.x. PMID 12190658
- [Background] Dizier MH, Besse-Schmittler C, Guilloud-Bataille M, Annesi-Maesano I, Boussaha M, Bousquet J, Charpin D, Degioanni A, Gormand F, Grimfeld A, Hochez J, Hyne G, Lockhart A, Luillier-Lacombe M, Matran R, Meunier F, Neukirch F, Pacheco Y, Parent V, Paty E, Pin I, Pison C, Scheinmann P, Thobie N, Vervloet D, Kauffmann F, Feingold J, Lathrop M, Demenais F. Genome screen for asthma and related phenotypes in the French EGEA study. Am J Respir Crit Care Med. 2000 Nov;162(5):1812-8. doi: 10.1164/ajrccm.162.5.2002113. PMID 11069818
- [Background] Xu W, Liu L, Emson PC, Harrington CR, Charles IG. Evolution of a homopurine-homopyrimidine pentanucleotide repeat sequence upstream of the human inducible nitric oxide synthase gene. Gene. 1997 Dec 19;204(1-2):165-70. doi: 10.1016/s0378-1119(97)00538-6. PMID 9434180
- [Background] Warpeha KM, Xu W, Liu L, Charles IG, Patterson CC, Ah-Fat F, Harding S, Hart PM, Chakravarthy U, Hughes AE. Genotyping and functional analysis of a polymorphic (CCTTT)(n) repeat of NOS2A in diabetic retinopathy. FASEB J. 1999 Oct;13(13):1825-32. doi: 10.1096/fasebj.13.13.1825. PMID 10506586
- [Background] Wildhaber JH, Hall GL, Stick SM. Measurements of exhaled nitric oxide with the single-breath technique and positive expiratory pressure in infants. Am J Respir Crit Care Med. 1999 Jan;159(1):74-8. doi: 10.1164/ajrccm.159.1.9805021. PMID 9872821
- [Background] Lundberg JO, Weitzberg E, Lundberg JM, Alving K. Nitric oxide in exhaled air. Eur Respir J. 1996 Dec;9(12):2671-80. doi: 10.1183/09031936.96.09122671. PMID 8980984
- [Background] George SC, Hogman M, Permutt S, Silkoff PE. Modeling pulmonary nitric oxide exchange. J Appl Physiol (1985). 2004 Mar;96(3):831-9. doi: 10.1152/japplphysiol.00950.2003. PMID 14766761
- [Background] Hamouda S, Chevalier-Bidaud B, Aboutaam R, Le Bourgeois M, Scheinmann P, Delclaux C, Mahut B. [Off-line exhaled nitric oxide measurement in children]. Rev Mal Respir. 2006 Nov;23(5 Pt 1):421-5. doi: 10.1016/s0761-8425(06)71811-3. French. PMID 17314740
- [Background] Mahut B, Louis B, Delclaux C. [Measurement of exhaled nitric oxide: methodology]. Rev Mal Respir. 2006 Jun;23(3 Suppl):6S29-6S36. French. PMID 16820746
- [Background] Paredi P, Loukides S, Ward S, Cramer D, Spicer M, Kharitonov SA, Barnes PJ. Exhalation flow and pressure-controlled reservoir collection of exhaled nitric oxide for remote and delayed analysis. Thorax. 1998 Sep;53(9):775-9. doi: 10.1136/thx.53.9.775. PMID 10319060
- [Background] Jobsis Q, Raatgeep HC, Hop WC, de Jongste JC. Controlled low flow off line sampling of exhaled nitric oxide in children. Thorax. 2001 Apr;56(4):285-9. doi: 10.1136/thorax.56.4.285. PMID 11254819
- [Background] Hall GL, Reinmann B, Wildhaber JH, Frey U. Tidal exhaled nitric oxide in healthy, unsedated newborn infants with prenatal tobacco exposure. J Appl Physiol (1985). 2002 Jan;92(1):59-66. doi: 10.1152/jappl.2002.92.1.59. PMID 11744643
- [Background] Gabriele C, van der Wiel EC, Nieuwhof EM, Moll HA, Merkus PJ, de Jongste JC. Methodological aspects of exhaled nitric oxide measurements in infants. Pediatr Allergy Immunol. 2007 Feb;18(1):36-41. doi: 10.1111/j.1399-3038.2006.00472.x. PMID 17295797
- [Background] Tabachnik E, Levison H. Postgraduate course presentation. Infantile bronchial asthma. J Allergy Clin Immunol. 1981 May;67(5):339-47. doi: 10.1016/0091-6749(81)90077-4. PMID 6785335
- [Background] Worldwide variation in prevalence of symptoms of asthma, allergic rhinoconjunctivitis, and atopic eczema: ISAAC. The International Study of Asthma and Allergies in Childhood (ISAAC) Steering Committee. Lancet. 1998 Apr 25;351(9111):1225-32. PMID 9643741
- [Background] Kauffmann F, Annesi-Maesano I, Liard R, Paty E, Faraldo B, Neukirch F, Dizier MH. [Construction and validation of a respiratory epidemiological questionnaire]. Rev Mal Respir. 2002 Jun;19(3):323-33. French. PMID 12166414
- [Background] Annesi-Maesano I, Didier A, Klossek M, Chanal I, Moreau D, Bousquet J. The score for allergic rhinitis (SFAR): a simple and valid assessment method in population studies. Allergy. 2002 Feb;57(2):107-14. doi: 10.1034/j.1398-9995.2002.1o3170.x. PMID 11929412
- [Background] Azevedo I, de Blic J, Scheinmann P, Vargaftig BB, Bachelet M. Enhanced arachidonic acid metabolism in alveolar macrophages from wheezy infants. Modulation by dexamethasone. Am J Respir Crit Care Med. 1995 Oct;152(4 Pt 1):1208-14. doi: 10.1164/ajrccm.152.4.7551372.